CLINICAL TRIAL: NCT02849977
Title: Genetic Testing and Phenotypic Characterization of Severely Obese Pediatric and Adult Volunteers
Status: Completed | Type: Observational
Sponsor: Rhythm Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: RM-493-013
Record Dates: First submitted 2016-07-26; First posted 2016-07-29 (Estimated); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Pro-opiomelanocortin (POMC), Proprotein Convertase Subtilisin/Kexin Type 1 (PCSK1) and Leptin Receptor (LepR) Gene Mutations
Keywords: POMC; PCSK1; Pro-opiomelanocortin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Cohort 1: If the subject has a history of hyperphagia, early onset obesity and/or clinical characteristics known to be related to mutations in the MC4R pathway and related to obesity (1.4 times 95th percentile in children).
- Cohort 2: If the subject has exponentially high BMI (≥50 to 59), without hyperphagia and early onset obesity, whose obesity may be driven by an MC4R pathway mutation in the absence of other clear history or clinical characteristics (1.5 - 1.6 times 95th percentile in children).
- Cohort 3: If the subject has exponentially high BMI (≥60), without hyperphagia and early onset obesity, whose obesity may be driven by an MC4R pathway mutation in the absence of other clear history or clinical characteristics (1.6 times 95th percentile in children).
- Cohort 4: If the subject has had or is undergoing bariatric surgery, who represents a refractory population of severely obese individuals whose obesity may be driven by an MC4R pathway mutation in the absence of other clear history or clinical characteristics (1.4 times 95th percentile in children and adolescents aged 12 and older).

SUMMARY:
The purpose of this screening study is to identify people who have a rare genetic cause of obesity - specifically three genetic variants (a change in the DNA structure) of the POMC, PCSK1 and LepR genes that are currently known to result in obesity.

This screening study will not include any investigational drugs. You will be asked to provide a DNA sample and answer some questions about your medical history and hunger.

ELIGIBILITY:
Individuals who meet any of the following inclusion criteria may be eligible:

1. Participant aged 2 or older.
2. Study participant and/or parent or guardian is able to communicate well with the investigator, to understand and comply with the requirements of the study, and be able to understand and sign the written informed consent/assent.
3. ≥40kg/m2 (age 18 and older) or 1.4x 95th percentile of BMI for age (ages 2-17) - with evidence of hunger or hyperphagia by screening surveys, indicated by a patient or observer score at or greater than midpoint of scale.

   o Individuals with clinical evidence of RGDO (per appendix 4) but do not meet the BMI criteria may be included if the investigators estimation and proband demonstrates a BMI Z-score difference of >1 between proband and any other sibling; and/or the proband demonstrates a BMI difference >10 kg/m2 between proband and parents.
4. ≥50 kg/m2 (age 18 and older) or 1.5x 95th percentile of BMI for age (ages 2-17). Cohorts included under this criteria include ≥50-60 kg/m2 (age 18 and older) or 1.5x 95th percentile of BMI for age (ages 2-17) and ≥60 kg/m2 (age 18 and older) or 1.6x 95th percentile of BMI for age (ages 2-17).
5. ≥ 40 kg/m2 (pre-operative) or 1.4x 95th percentile of BMI for age (ages 12-17) with history of bariatric surgery or planned surgery within 3 months (prior to or following screening).

Individuals who meet any of the following exclusion criteria will not be eligible:

1. Prior craniopharyngioma or other hypothalamic brain region surgery or surgeries/procedures for brain tumor, i.e., ventriculoperitoneal shunt and radiation therapy
2. Diagnosis of Prader-Willi syndrome

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The objective is to identify individuals with severe, early onset morbid obesity (EOMO), who are aged 2 years of age or older, and are suspected to be either homozygous, compound heterozygous or heterozygous for loss of function mutations in the POMC, PCSK1 or LepR gene, leading to a clinical presentation of Melanocortin 4 (MC4) pathway deficiency obesity. Individuals may be contacted for further assessment of clinical features (including questionnaires on past weight and medical history and current hunger and feeding behavior symptoms) and/or participation in future Rhythm clinical trials.
Sampling Method: Non-Probability Sample
Enrollment: 5966 (Actual)
Dates: Start 2016-09-28 (Actual); Primary Completion 2020-06-09 (Actual); Study Completion 2020-06-09 (Actual)

PRIMARY OUTCOMES:
Identification of individuals with POMC, LepR or PCSK1 genetic mutations | 1 Year

CONTACTS AND LOCATIONS:
Overall Officials: David Meeker, Study Chair — Rhythm Pharmceuticals, Inc.
Locations (58):
- United States (48):
  - Synexus Clinical Research US, Inc. - Simon Williamson Clinic, PC, Birmingham, Alabama
  - Synexus Clinical Research US, Inc. - Phoenix Southeast, Chandler, Arizona
  - Clinical Research Advantage Inc., Mesa, Arizona
  - Tucson Neuroscience Research - M3 Wake Research, Tucson, Arizona
  - Encino, California
  - PRI, LLC - Los Alamitos - M3 Wake Research, Los Alamitos, California
  - Axis Clinical Trails, Los Angeles, California
  - Axis Clinical Trials, Los Angeles, California
  - PRI, LLC - Newport Beach - M3 Wake Research, Newport Beach, California
  - Nemours Foundation Alfred Dupont Children's Hospital, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Florida, Gainesville, Florida
  - South Florida Clinical Trials, Hialeah, Florida
  - Translational Research Inst. for Metabolism and Diabetes, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Palm Harbor Medical Associates - BTC - PPDS, Palm Harbor, Florida
  - Synexus Clinical Research US, Inc. - St. Petersburg, Pinellas Park, Florida
  - Synexus Clinical Research US, Inc. - Chicago, Chicago, Illinois
  - Maine Medical Partners Pediatric Specialty Care, Portland, Maine
  - Baystate Children's Hospital, Division of Pediatric Endocrinology, Springfield, Massachusetts
  - Helen DeVos Children's Hospital Healthy Weight Center, Grand Rapids, Michigan
  - Synexus Clinical Research US, Inc. - West Florissant Internists, Bridgeton, Missouri
  - Impact Clinical Trials - Las Vegas, Las Vegas, Nevada
  - University of New Mexico, Albuquerque, New Mexico
  - New York Clinical Trials-Brooklyn, Brooklyn, New York
  - Division of Endocrinology/Diabetes Amanda House, Buffalo, New York
  - Cohen Children's Medical Center of NY, Lake Success, New York
  - NYU Langone Medical Center, New York, New York
  - Columbia University, New York, New York
  - New York Clinical Trials-Manhattan, New York, New York
  - UNC Health Care - NC Children's Specialty Clinic, Chapel Hill, North Carolina
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke University Hospital, Durham, North Carolina
  - Synexus Clinical Research US, Inc. - Akron, Akron, Ohio
  - Synexus Clinical Research US, Inc. - Cincinnati, Cincinnati, Ohio
  - Nationwide Children's Hospital, Center for Healthy Weight and Nutrition, Columbus, Ohio
  - Synexus Clinical Research US, Inc. - Columbus, Columbus, Ohio
  - Synexus Clinical Research US, Inc. - Centennial Health, PC -, Oklahoma City, Oklahoma
  - Synexus Clinical Research US, Inc. - Primary Care Associates, Anderson, South Carolina
  - University of Tennesseee Health Science Center, Memphis, Tennessee
  - Medical Research Center of Memphis, LLC - M3 Wake Research, Memphis, Tennessee
  - Vanderbilt University, Nashville, Tennessee
  - Texas Tech University Health Sciences Center, Amarillo, Texas
  - Synexus - Synexus US, LP - Dallas, Dallas, Texas
  - Global Medical Research - M3 Wake Research, DeSoto, Texas
  - Synexus Clinical Research US, Inc. - San Antonio, San Antonio, Texas
  - University of Utah, Department of Surgery, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington
- University of Alberta, Edmonton, Alberta, Canada
- Charite Campus Virchow-Klinikum Institute for Experimental Pediatric Endocrinology, Berlin, Germany
- University of Hospital of Patras, Pátrai, Greece
- Israel (5):
  - Rabin Medical Center - PPDS, Petah Tikva
  - Schneider Children's Medical Center of Israel - Petah Tikvah - PIN, Petah Tikva
  - Chaim Sheba Medical Center, Ramat Gan
  - Kaplan Medical Center, Rehovot
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- IRCCS Istituto Auxologico Italiano, Oggebbio, Italy
- Hospital Senhora da Oliveira -Guimaraes, E.P.E, Guimarães, Portugal

IPD SHARING:
Plan to Share IPD: No